CLINICAL TRIAL: NCT06028256
Title: Continuous Norepinephrine Infusion Before General Anesthesia to Prevent Post-induction Hypotension in High-risk Patients Undergoing Major Noncardiac Surgery
Brief Title: Norepinephrine Prevent Post-induction Hypotension in High-risk Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yuan Chang, Principal Investigator, First Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-L-126
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia; Blood Pressure; Norepinephrine
Keywords: intraoperative hypotension; arterial pressure; general surgery; general anesthesia; noncardiac surgery
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine (Experimental): The interventional group will receive a continuous infusion of norepinephrine 5 minutes (0.01μg/kg*min) before anesthesia induction until skin incision.
  Interventions: Drug: Norepinephrine Hydrochloride
- Placebo (Placebo Comparator): the placebo group will receive a continuous infusion of normal saline (10 ml/h) 5 minutes before anesthesia induction until skin incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norepinephrine Hydrochloride — Both arms of patients will receive standard anesthesia and surgical management. Radial artery cannulation and invasive blood pressure monitoring will be perform.
  Norepinephrine will be pumped at a rate of 10 ml/h for 5 minutes before anesthesia induction to skin incision.
  Arms: Norepinephrine
Drug: Placebo — Normal saline will be pumped at a rate of 10 ml/h for 5 minutes before anesthesia induction to skin incision.
  Arms: Placebo

SUMMARY:
The investigators aimed to investigate the effects of continuous infusion of norepinephrine before and after general anesthesia induction on the occurrence of post-induction hypotension.

DETAILED DESCRIPTION:
Intraoperative hypotension is common after general anesthesia induction and is associated with adverse postoperative events. Norepinephrine is one of the most applied vasopressors in clinical to treat intraoperative hypotension. Due to the absence of effective measures for predicting intraoperative hypotension, infusing norepinephrine before and during anesthesia induction may reduce intraoperative hypotension. There is currently a lack of research regarding whether continuous norepinephrine infusion before and during the induction of general anesthesia can mitigate or prevent post-induction hypotension. The investigators aim to investigate the effects of continuous infusion of norepinephrine before and after general anesthesia induction on the occurrence of post-induction hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 65 years or those above 45 years with at least one of the following preoperative cardiovascular diseases: essential hypertension, coronary artery disease, stroke, or type I/II diabetes mellitus.
* Patients who will receive major noncardiac surgery as open or laparoscopic abdominal surgeries with an anticipated operative duration over two hours, including gastrointestinal, liver, pancreatic, bladder, and uterine/adnexal surgeries.

Exclusion Criteria:

* Patients who declined to participate in the present study.
* Patients enrolled in another ongoing clinical study.
* Patients with systolic arterial pressure (SAP) below 90 mmHg or above 160 mmHg, or heart rate (HR) over 100 beats per minute (bpm) before anesthesia induction.
* Patients who have experienced any type of shock within 30 days before surgery.
* Patients with circulatory instability require continuous or intermittent positive inotropic and/or vasopressors within 24 hours before surgery.
* Patients receive continuous or intermittent intravenous antihypertensive agents within 24 hours before surgery.
* Patients underwent coronary artery bypass grafting, coronary angiography, or coronary stenting within 180 days before surgery.
* Patients who were diagnosed with new-onset tachyarrhythmia within 180 days before surgery, such as atrial fibrillation, atrial flutter, and premature ventricular contractions.
* Patients with preoperative alanine aminotransferase >80 international units and/or glomerular filtration rate < 80 ml/min within the 180 days before surgery.
* Patients are ineligible for intraoperative invasive radial artery blood pressure monitoring.
* Patients with a known history of allergy to norepinephrine.
* Patients who were planned for rapid sequence induction.
* Patients who were scheduled for awake tracheal intubation.
* Patients who were scheduled for double-lumen endotracheal intubation. Pregnant or lactating patients.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-induction hypotension | From induction of general anesthesia to skin incision (up to one hour from induction of general anesthesia)
  Hypotension: mean arterial pressure (MAP) <65 mmHg

SECONDARY OUTCOMES:
Incidence of the following abnormal vital signs | From induction of general anesthesia to skin incision (up to one hours from induction of general anesthesia)
  MAP<65 mmHg, MAP<55 mmHg, MAP decreased over 20% ,30% and 40% from preoperative level; MAP increased over 20%, 30%, and 40% from preoperative level; SAP < 90 mmHg; Systolic arterial pressure (SAP) > 160 mmHg; Heart rate (HR) < 40 bpm, HR > 100 bpm; dosage of norepinephrine given by anesthesiologists; amount of fluid; the time-point of the first events of MAP < 65 mmHg, MAP < 55 mmHg, SAP < 90 mmHg, SAP > 160 mmHg, MAP increased over 20%, 30%, and 40% from preoperative level.
Incidence of the following abnormal vital signs | From surgical incision to the end of surgery (up to six hours from surgical incision)
  MAP<65 mmHg, MAP<55 mmHg, MAP decreased over 20%, 30%, and 40% from preoperative level; MAP increased over 20%, 30%, and 40% from preoperative level; SAP < 90 mmHg; SAP > 160 mmHg; HR < 40 bpm, HR > 100 bpm. Dosage of norepinephrine given by anesthesiologists; amount of fluid; the time-point of the first events of MAP < 65 mmHg, MAP < 55 mmHg, SAP < 90 mmHg, SAP > 160 mmHg, MAP increased over 20%, 30%, and 40% from preoperative level
Incidence of the following abnormal vital signs | from the end of surgery until leaving the post-anesthesia care unit (up to four hours from the end of surgery)
  MAP<65 mmHg, MAP<55 mmHg, MAP decreased over 20%, 30%, and 40% from preoperative level; MAP increased over 20%, 30%, and 40% from preoperative level; SAP < 90 mmHg; SAP > 160 mmHg; HR < 40 bpm, HR > 100 bpm. Dosage of norepinephrine given by anesthesiologists; amount of fluid; the time-point of the first events of MAP < 65 mmHg, MAP < 55 mmHg, SAP < 90 mmHg, SAP > 160 mmHg, MAP increased over 20%, 30%, and 40% from preoperative level
Postoperative major adverse cardiac events | Within 30 days after surgery
  Cardiac death, myocardial infarction, on-fatal cardiac arrest, coronary revascularization

IPD SHARING:
Plan to Share IPD: No